CLINICAL TRIAL: NCT05838326
Title: Physiological Effects of High Flow Oxygen Therapy Using 'Optiflow + Duet' Interface vs 'Standard' High Flow Nasal Cannula for Acute Respiratory Failure After Extubation. The OPTIMARF Study.
Brief Title: 'Optiflow + Duet' Interface' vs 'Standard' High Flow Nasal Cannula
Acronym: OPTIMARF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AOP2949
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Hypoxemia
Keywords: asymmetrical nasal cannula; hypoxemia; DUET
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symmetrical high flow nasal cannula (HFNO) (Active Comparator): After a 'baseline' trial using Venturi Mask, within the first 120 minutes after extubation, and assessing a arterial oxygen pressure (PaO2) and inspiratory oxygen fraction (FiO2) ratio < 300, patients will be randomly assigned to a first 1h-phase of 'conventional HFNO' or 'DUET HFNO'. At the end of each session several clinical parameters (i.e. DUS, EIT, ABGs, comfort, VAS) will be collected.
  Specifically, Gas-flow rate will be set at a maximum of 60 L/min, temperature at a maximum of 37°C, while FiO2 will be adjusted to maintain a peripheral saturation (SpO2) between 92 and 98%.
  Interventions: Device: Symmetrical high flow nasal cannula (HFNO)
- Asymmetrical high flow nasal cannula (DUET HFNO) (Active Comparator): After a 'baseline' trial using Venturi Mask, within the first 120 minutes after extubation, and assessing a PaO2/FiO2 ratio < 300 (as described above), patients will be randomly assigned to a second 1h-phase of 'DUET HFNO' vs 'conventional HFNO'. At the end of each session several clinical parameters (i.e. DUS, EIT, ABGs, comfort, VAS) will be collected.
  Specifically, Gas-flow rate will be set at a maximum of 60L/min, temperature at a maximum of 37°C, while FiO2 will be adjusted to maintain SpO2 between 92 and 98%.
  Interventions: Device: Asymmetrical high flow nasal cannula (DUET HFNO)

INTERVENTIONS:
Device: Symmetrical high flow nasal cannula (HFNO) — After a 'baseline' trial using Venturi Mask, within the first 120 minutes after extubation, and assessing a PaO2/FiO2 ratio < 300, patients will be randomly assigned to a first 1h-phase of 'conventional HFNO' or 'DUET HFNO'. At the end of each session several clinical parameters (i.e. DUS, EIT, ABGs, comfort, VAS) will be collected.
  Specifically, Gas-flow rate will be set at a maximum of 60 L/min, temperature at a maximum of 37°C, while FiO2 will be adjusted to maintain SpO2 between 92 and 98%.
  Arms: Symmetrical high flow nasal cannula (HFNO)
Device: Asymmetrical high flow nasal cannula (DUET HFNO) — After a 'baseline' trial using Venturi Mask, within the first 120 minutes after extubation, and assessing a PaO2/FiO2 ratio < 300, patients will be randomly assigned to a first 1h-phase of 'DUET HFNO' vs 'conventional HFNO'. At the end of each session several clinical parameters (i.e. DUS, EIT, ABGs, comfort, VAS) will be collected.
  Specifically, Gas-flow rate will be set at a maximum of 60 L/min, temperature at a maximum of 37°C, while FiO2 will be adjusted to maintain SpO2 between 92 and 98%.
  A 5-10min 'washout' phase using VM, between different interfaces, will be allowed.
  Arms: Asymmetrical high flow nasal cannula (DUET HFNO)

SUMMARY:
High-flow nasal cannula (HFNC) therapy is increasingly used in the management of acute respiratory failure. Its clinical application has been largely investigated in chronic obstructive pulmonary disease (COPD) patients but only marginally in patients experiencing acute respiratory failure after extubation. Promising data have been published in vitro about new asymmetrical high flow nasal cannula, named 'Optiflow + DUET'. Positive airway pressure, that dynamically changes with breathing, and clearance of anatomical dead space are the key mechanisms of noninvasive respiratory support with nasal high flow. Pressure mainly depends on flow rate and nare occlusion. The hypothesis is that an increase in asymmetrical occlusion of the nares leads to an improvement in dead-space clearance resulting in a reduction in re-breathing and breathing work.

DETAILED DESCRIPTION:
A prospective cross-over RCT on the effects of 'Optiflow + DUET' as compared to convetional symmetrical high flow cannula and Venturi mask.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old;
* invasive mechanical ventilation > 24h;
* acute respiratory failure within 120 minutes after extubation (defined during a spontaneous trial using Venturi mask and assessing a PaO2/FiO2 ratio < 300;
* absence of Sars-Cov-2 positivity;
* absence of cardiological or long-term respiratory disease

Exclusion Criteria:

* pregnancy
* tracheostomy
* non-invasive ventilation after extubation
* second tracheal intubation
* contraindications for EIT belt
* facial or nose abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Breathing effort | Last 10 minutes of 1 hour-trial
  To evaluate changes, between arms, in breathing effort (as assessed by diaphragm ultrasound (DUS)).
Lung aeration | Last 10 minutes of 1 hour-trial
  To evaluate changes, between arms, in lung aeration (as assessed by the end-expiratory lung impedance (delta EELI) through EIT.

SECONDARY OUTCOMES:
Minute ventilation (MV) (L/min) | Last 10 minutes of 1 hour-trial
  To evaluate breathing pattern
corrected MV (L/min) | Last 10 minutes of 1 hour-trial
  To evaluate breathing pattern
Breathing heterogeneity | Last 10 minutes of 1 hour-trial
  To evaluate changes, between arms, in ventilation distribution (as assessed by pendelluft (yes/not), respiratory rates/min, tidal volume (ml), global inhomogeneity index through EIT)
Comfort | Last 10 minutes of 1h-trial
  To evaluate changes in comfort, between arms, as assessed by NRS scale
Dyspnea | Last 10 minutes of 1h-trial
  To evaluate changes in dyspnea, between arms, as assessed by VAS scale
Gas exchange | Last 10 minutes of 1h-trial
  To evaluate changes, between arms, in gas exchange (as assessed by PaO2 mmHg, pCO2 mmHg, pH through ABGs)

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Boscolo, MD, Principal Investigator — AOUP, DIMED
Locations (1):
- Institute of Anaesthesia and Intensive Care, Padua University hospital, Padua, Italy

REFERENCES:
- [Derived] Boscolo A, Pettenuzzo T, Zarantonello F, Sella N, Pistollato E, De Cassai A, Congedi S, Paiusco I, Bertoldo G, Crociani S, Toma F, Mormando G, Lorenzoni G, Gregori D, Navalesi P. Asymmetrical high-flow nasal cannula performs similarly to standard interface in patients with acute hypoxemic post-extubation respiratory failure: a pilot study. BMC Pulm Med. 2024 Jan 8;24(1):21. doi: 10.1186/s12890-023-02820-x. PMID 38191347